CLINICAL TRIAL: NCT06147245
Title: A Person-centred and Culturally Sensitive Course of Treatment Targeting Individuals With Type 2 Diabetes and Non-Western Backgrounds (The ACCT2 Study)
Brief Title: The ACCT2 Study Individuals With Type 2 Diabetes and Non-Western Backgrounds (ACCT2)
Acronym: ACCT2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23042245
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Glycaemic control; Cultural Sensitivity; Diabetes self-management; Non-Western immigrants; Co-creation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Person-centred culturally sensitive course of treatment (Experimental): The intervention consists of a 12-month person-centred and culturally sensitive course of treatment.
  Interventions: Behavioral: Person-centred culturally sensitive course of treatment
- Control (No Intervention): The control group will follow the standard care with regular visits at the T2D outpatient clinic at SDCC 3-4 times/year.

INTERVENTIONS:
Behavioral: Person-centred culturally sensitive course of treatment — 12-month person-centred and culturally sensitive intervention: Participants will attend 6 visits at SDCC including visits with a diabetes nurse, physician and dietitian. The course of treatment is focusing on extended time in consultations, use of technology for diabetes monitoring, meeting the same healthcare professionals, awareness of language barriers and use of accurate communication and dialogue tools in participants native language.
  Arms: Person-centred culturally sensitive course of treatment

SUMMARY:
The overall purpose of the present study is to examine the effect of implementing a 12-month person-centred and culturally sensitive intervention on glycaemic control in individuals with type 2 diabetes (T2D) and a non-Western background. We hypothesise that the intervention added to standard care will be superior for reducing HbA1c. Superiority will be claimed if the baseline corrected difference between the two groups is equal to, or surpass, the minimal important difference (5 mmol/mol) in favour of the intervention-group.

DETAILED DESCRIPTION:
Individuals with a non-Western background have a higher prevalence of T2D and exhibit poorer glycaemic control (HbA1c levels) than those with Danish ethnic background. Research indicates that individuals with non-Western backgrounds face a number of challenges for effective diabetes management. These challenges include low health literacy, language barriers in accessing and comprehending information, adherence to medication, lifestyle factors, and limited social support. Although studies show that culturally appropriate diabetes education can enhance glycaemic control and improve health behaviours, little is known about effective strategies and methods targeting individuals with non-Western backgrounds and T2D. This suggests a strengthened and systematic effort towards the treatment of individuals with T2D and non-Western backgrounds.

Overall, the ACCT2 study consists of three phases; 1) Need assessment, 2) Intervention development and testing, and 3) Randomized controlled trial (RCT). The aim of the present study (RCT) is to examine the effectiveness of a 12-month person-centred and culturally sensitive intervention on glycaemic control in individuals with T2D and a non-Western background (speaking either Urdu, Arabic or Turkish as native language). Participants will attend 6 visits at Steno Diabetes Center Copenhagen (SDCC): Visit 1 (baseline), visit 2 (two weeks after baseline), visit 3 (4 weeks after baseline), visit 4 (4 months after baseline), visit 5 (7-8 months after baseline), visit 6 (12 months after baseline).

The specific objectives are:

1. To investigate the effect of a 1-year person-centred and culturally sensitive intervention on change in glycaemic control (HbA1c)
2. To describe changes in cardiometabolic risk factors (including blood lipids, markers of glucose metabolism, blood pressure)
3. To describe changes in patient-reported outcomes including overall health, well-being, quality of life, social support, diabetes management, diabetes distress, health behaviour, health literacy, medicine adherence, time-below-range (TBR), time-above-range (TAB), time-in-range (TIR), body weight and use of antidiabetic medicine
4. To describe the extent to which the intervention was conducted as planned (visits, person-centred approach, tools)
5. To explore participants' experiences with following the intervention and acceptance of it, including how a person-centred and culturally sensitive approach worked for them as well as the use of using technology for diabetes monitoring (sub-population).

ELIGIBILITY:
Inclusion Criteria:

* Having T2D with poor glycaemic control (HbA1c ≥53 mmol/mol) and where individual treatment goal for HbA1c has not been achieved (in two consecutive measurements)
* Having a non-Western background speaking either Urdu, Arabic or Turkish as native language
* Already in a course of treatment at the outpatient T2D clinic at SDCC

Exclusion Criteria:

* Age: > 75 years
* Residing part-time in Denmark
* Marker of kidney function - estimated glomerular filtration rate (eGFR) below 30 mL/min
* Having severe mental disorders
* Having disabilities inhibiting physical attendance
* Participant's general condition contraindicates continuing the study, as judged by the investigator or a medical expert
* Participant's withdrawal of the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (mmol/mol) | Change from baseline to the end of intervention (12 months)
  Assessed from blood samples in non-fasted state

SECONDARY OUTCOMES:
Blood lipids (mmol/l) | Change from baseline to the end of intervention (12 months)
  Concentrations of: Total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides
Systolic blood pressure (mmHg) | Change from baseline to the end of intervention (12 months)
  Measured in resting state. Blood pressure measurements are repeated three times and mean value is calculated
Diastolic blood pressure (mmHg) | Change from baseline to the end of intervention (12 months)
  Measured in resting state. Blood pressure measurements are repeated three times and mean value is calculated
Resting heart rate (bpm) | Change from baseline to the end of intervention (12 months)
  Measured in resting state
Marker of kidney function - Creatinine (μmmol/L) | Change from baseline to the end of intervention (12 months)
  Concentration of creatinine
Marker of kidney function - eGFR (mL/min) | Change from baseline to the end of intervention (12 months)
  Estimated glomerular filtration rate (eGFR)
Serum sodium (mmol/L) | Change from baseline to the end of intervention (12 months)
  Serum sodium concentration
Serum potassium (mmol/L) | Change from baseline to the end of intervention (12 months)
  Serum potassium concentration
Thyroid-stimulating hormone (TSH) (mIU/L) | Change from baseline to the end of intervention (12 months)
  Level of TSH assessed from blood samples
Marker of liver function - Alanine aminotransferase (U/L) | Change from baseline to the end of intervention (12 months)
  Concentration of alanine aminotransferase
C-peptide | Change from baseline to the end of intervention (12 months)
  Plasma concentration of c-peptide
Coefficient of variation (CV) of glucose concentrations | Change from baseline to the end of intervention (12 months)
  Measured using continous glucose monitoring
Screening for diabetic nephropathy - Urine albumin (mg)/creatinine (g) ratio | Change from baseline to the end of intervention (12 months)
  Measured in a urine sample

OTHER OUTCOMES:
Time-in-range (% 3.9-10.0 mmol/l) | Change from baseline to the end of intervention (12 months)
  Measured using continous glucose monitoring
Time-below-range (% <3.9 mmol/l) | Change from baseline to the end of intervention (12 months)
  Measured using continous glucose monitoring
Time-above-range (% >10.0 mmol/l) | Change from baseline to the end of intervention (12 months)
  Measured using continous glucose monitoring
Body weight (kg) | Change from baseline to the end of intervention (12 months)
  Measured on a digital scale
Use of antidiabetic medication | Change from baseline to the end of intervention (12 months)
  Change in current use of antidiabetic medication
Self-reported well-being | Change from baseline to the end of intervention (12 months)
  Assessed from the WHO-5 well-being index.The WHO-5 consists of five statements, which respondents rate from 0 to 5 (in relation to the past two weeks).The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being
Self-reported diabetes distress | Change from baseline to the end of intervention (12 months)
  Assessed from the Problem Areas in Diabetes Scale (PAID-5 scale) comprising five of the emotional-distress questions of the full PAID items. Each item can be rated from 0 to 4. A total score of ≥ 8 indicates possible diabetes related emotional distress.
Self-reported diabetes management | Change from baseline to the end of intervention (12 months)
  Assessed from 9 selected items on diabetes management from The Danish National Patient Reported Outcome Questionnaire (Danish PRO scheme (diabetes), item 27-35). The items can be rated from 'very sure/confident' to 'not sure/confident at all'.
Self-reported information regarding social support | Change from baseline to the end of intervention (12 months)
  Assessed from item 70 of social support questionnaire (the Danish National Health Survey, item 70). The question refers to contact with other people.
Medicine adherence | Change from baseline to the end of intervention (12 months)
  Assessed from the MARS-5. The questions can be rated from 1 to 5. The MARS-5 score is calculated by summing the numeric score (range 1-5) from each question. A higher score indicates better adherence.
Health literacy | Change from baseline to the end of intervention (12 months)
  Assessed from 3 selected items from the Health Literacy Questionnaire (HLQ).
Degree of participants' participation in intervention activities | There are 6 visits overall and participation will be measured at the end of the intervention (12 months after baseline).
  Assessed from % participation in visits
Participants' acceptance of intervention | The interviews will be conducted at the end of intervention (12 months after baseline) at visit 6.
  Assessed by individual interviews on participants' acceptance of intervention in terms of experiences and how intervention activities were supportive. This refers only to the intervention group. Individual interviews will be conducted by a qualitative researcher with a sub-group of participants in the intervention group after the last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Bjerre-Christensen, MD, Principal Investigator — Steno Diabetes Center Copenhagen; Natasja B Martinsen, PhD, Study Director — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

REFERENCES:
- [Derived] Bjerre N, Christensen L, Hoeiberg C, Ottosson C, Jensen MK, Kildsig N, Moller TK, Termannsen AD, Ewers B, Hollender-Schou B, Grue RM, Bjerre-Christensen U, Jansen S, Akram K. Effectiveness of a Person-Centered and Culturally Sensitive Course of Treatment in Arabic-, Turkish-, and Urdu-Speaking Individuals With Type 2 Diabetes (the ACCT2 Study): Protocol for a Pragmatic Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 5;14:e67319. doi: 10.2196/67319. PMID 40471662